CLINICAL TRIAL: NCT06500533
Title: Combined rTMS/tDCS in Unipolar Depression: an Exploratory Open-label Trial
Brief Title: Combining rTMS and tDCS in Depression: an Exploratory Clinical Trial
Acronym: CombTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principal Investigator left the institution, resulting in the inability to maintain necessary conditions for study continuation. Sufficient data were collected for scientific analysis, but not all planned data were obtained.
Sponsor: Regionspsykiatrien Gødstrup (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Open label TMS
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Major Depression; Treatment Resistant Depression
Keywords: unipolar depression; rTMS; tDCS; neuromodulation; treatment resistant depression; difficult-to-treat depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depressive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study's single arm (Experimental): Patients will be receiving rTMS/tDCS combined 30-session protocol, consisting of 15 rTMS sessions every other day alternating with 15 tDCS at-home treatments.
  The rTMS protocol used in the study will be intermittent Theta Burst Stimulation (iTBS) on the left dorsolateral prefrontal cortex given for 3 minutes and 9 seconds, every other day 5 weeks. iTBS is delivered in 2s bursts consisting of three pulses at a frequency of 50 Hz, with an inter-burst interval of 200 ms (i.e., 5 Hz). Stimulation intensity will be 120% of resting motor threshold.
  Each of the 15 tDCS sessions will be lasting 30 minutes with a stimulation intensity of 2mA. The electrodes will be positioned bilaterally over the dorsolateral prefrontal cortex. The device chosen for the study is specifically designed for home use. The device is controlled via an app that walks the participant through correct usage and dosage with the device to minimize non-compliance.
  Interventions: Device: rTMS combined with tDCS

INTERVENTIONS:
Device: rTMS combined with tDCS — The intervention will last 30 days per patient, where rTMS will be administered on odd numbered days (study day 1, 3, 5, 7, ..29) and tDCS on even numbered days (study day 2, 4, 6, 8, … 30). All patients will start with TMS and finish with home-based tDCS treatment. Both rTMS and tDCS treatments will be administered during working days, from Monday to Friday.
  rTMS treatment will be administered by the experienced nurses of the rTMS clinic of each department. The rTMS treatment will profit from ongoing supervision by the Clinical Directors of each TMS clinic, which is in line with treatment as usual.
  tDCS will be performed at home by the patients.

SUMMARY:
The investigators aim to conduct a single-arm open-label clinical trial, meaning that the investigators will be administering a treatment protocol to one group of patients, where no information is withheld from trial participants.

The treatment being researched will consist of a rTMS/tDCS combined 30-session protocol, consisting of 15 rTMS sessions every other day alternating with 15 tDCS at-home treatments. Treatment sessions will occur from Monday to Friday.

rTMS (Repetitive Transcranial Magnetic Stimulation) is a non-invasive physical treatment, which uses pulsing magnetic fields to activate or suppress the brain centres associated with medical and psychiatric disorders, thus treating the brain circuits involved in the patient's condition. tDCS (transcranial direct current stimulation) is a form of neuromodulation that uses constant, low direct current delivered via electrodes on the head.

The investigators aim to recruit 40 patients with difficult to treat unipolar depression. Patients will be selected among the referrals to the psychiatry department in Gødstrup and to the psychiatry department in Randers.

rTMS treatment will be administered by the experienced nurses of the rTMS clinic of each department. The TMS treatment will profit from ongoing supervision by the Clinical Directors of each rTMS clinic. tDCS will be performed at home by the patients.

The study itself will last 30 days per patient, where rTMS will be administered on odd numbered days (study day 1, 3, 5, 7, ..29) and tDCS on even numbered days (study day 2, 4, 6, 8, … 30). All patients will start with rTMS and finish with home-based tDCS treatment. Both rTMS and tDCS treatments will be administered during working days, from Monday to Friday. The trial itself is expected to last no more than two years.

The goal of this study then is to examine the effectiveness of this combined neuromodulation intervention, which has the advantage of reducing the attendance requirements for TMS treatment by 50%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 22 and 80 years of age.
* Able to provide informed consent.
* Primary diagnosis of depressive episode (F32) or recurrent depressive disorder (F33), according to International Classification of Diseases 10th Revision (ICD-10).
* Simultaneous fulfillment of diagnostic criteria for Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE), according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Currently experiencing moderate to severe depressive episodes (scores ≥20 on the 17-item Hamilton Depression Rating Scale [HAM-D 17]).

Exclusion Criteria:

* Primary psychiatric diagnosis other than single episode depressive disorder or recurrent depressive disorder.
* History of schizophrenia or schizoaffective disorders.
* Any history of psychotic symptoms in the current or previous depressive episodes.
* History of obsessive-compulsive disorder.
* History of autism spectrum disorder.
* History of intractable migraine.
* Clinical conditions that would increase risks associated with receiving high-dose iTBS.
* Cochlear implants.
* Epilepsy.
* Pacemakers.
* Presence of metal in the head, especially of a ferromagnetic type.
* Presence of magnetically controlled implantable devices.
* Current drug misuse (F10-F19).
* History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
* Current (or chronic) use of opiates.
* Prior nonresponse to rTMS.
* Prior nonresponse to Electroconvulsive Therapy (ECT).
* Female that is pregnant or breastfeeding.
* Female with a positive pregnancy test at participation.
* History of psychosurgery for depression.
* Damage to- or diseases of the skin, which affects the scalp. E.g. Psoriasis or open wounds.
* No changes in psychotropic medication during the study will be allowed, with the exception of the ones due to intolerability.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
HAM-D17 scores | Baseline, and end of the 30th treatment session.
  Our primary outcome measure will be Hamilton Depression Rating Scale, 17-item version (HAM-D17) scores at the end of the 30th treatment session normalized to baseline.

SECONDARY OUTCOMES:
HAM-D17 scores at week 9 and MDI scores | Baseline, end of the 30th treatment session and 4 weeks after the last treatment.
  Changes in HAM-D17 scores from baseline to 4 weeks after the last treatment (study week 9) will be a secondary outcome.
  HAM-D17 scores will be used to calculate response and remission rates in each group:
  * Response: reduction ≥50% in HAM-D17
  * Remission: HAM-D17 scores ≤7
  Our secondary outcome will also include changes in scores on the MDI will be used as a secondary measure of depression severity (30th session; 4 weeks after the 30th session), normalized to baseline. MDI scores will be used to calculate response and remission rates in each group:
  * Response: reduction ≥50% in MDI
  * Remission: MDI scores ≤20
  Response and remission at a single time point
  * Participants will be identified as responders or remitters if they met these specific criteria at day 30.
  * Participants will be identified as long-term responders or remitters if they meet these specific criteria at both study day 30 and study week 9 (e.g., 4 weeks after the end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro C Barata, MD, Principal Investigator — Regionspsykiatrien Gødstrup
Locations (1):
- Regionspsykiatrien Gødstrup, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No